CLINICAL TRIAL: NCT03807024
Title: Age-specific Prevalence and Comparisons of Urodynamics and Bladder Diary Between Overactive Bladder-wet and -Dry Women Based on Bladder Diary
Brief Title: Age-specific Prevalence and Comparisons of UDS and Bladder Diary Between OAB-wet and -Dry Women
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201810084RIND
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-12

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder; Bladder diary
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OAB-wet: The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The presence of at least one episode of urgency associated incontinence was defined to be OAB-wet.
  Interventions: Diagnostic Test: Bladder diary
- OAB-dry: The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The absence of urgency associated incontinence was defined to be OAB-dry.
  Interventions: Diagnostic Test: Bladder diary

INTERVENTIONS:
Diagnostic Test: Bladder diary — 3-day bladder diary: The classification of OAB-wet or OAB-dry is based on the record of the three-day bladder diary of each patient. The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The presence of at least one episode of urgency associated incontinence was defined to be OAB-wet, otherwise, OAB-dry
  Other Names: Questionnaire; Urodynamic study; Pad test

SUMMARY:
The knowledge of the age-specific prevalence of overactive bladder syndrome (OAB)-wet and -dry women is important for understanding the impact of aging on OAB. Thus, our aim is to describe clinically differences between OAB-wet and -dry women.

DETAILED DESCRIPTION:
Between July 2009 and January 2018, all women with OAB visiting a medical center for evaluation were reviewed. The classification of OAB-wet or OAB-dry is based on the record of the three-day bladder diary of each patient. The diagnosis of OAB in each patient was based on the presence of at least one episode of urgency in her three-day bladder diary and with the absence of stress urinary incontinence. The presence of at least one episode of urgency associated incontinence was defined to be OAB-wet, otherwise, OAB-dry.

ELIGIBILITY:
Inclusion Criteria:

1. More than 20-year-old
2. Female
3. Diagnosed with overactive bladder by bladder diary

Exclusion Criteria:

1. Younger than 20-year-old
2. Pregnant or planned to be pregnant

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2009 and January 2018, all women older than 20-year-old with OAB visiting a medical center for evaluation were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1071 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of OAB | Between July 2009 and January 2018
  Diagnosis of OAB according to ICS terminology guideline: Urgency, with or without urge incontinence, usually with frequency and nocturia, can be described as the overactive bladder syndrome, urge syndrome or urgency-frequency syndrome

SECONDARY OUTCOMES:
Age-specific comparison | Between July 2009 and January 2018
  Use questionnaire and urodynamic study to evaluate if there is difference between OAB-wet and OAB-dry women

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Powell LC, Szabo SM, Walker D, Gooch K. The economic burden of overactive bladder in the United States: A systematic literature review. Neurourol Urodyn. 2018 Apr;37(4):1241-1249. doi: 10.1002/nau.23477. Epub 2018 Jan 13. PMID 29331047
- [Background] Coyne KS, Wein A, Nicholson S, Kvasz M, Chen CI, Milsom I. Economic burden of urgency urinary incontinence in the United States: a systematic review. J Manag Care Pharm. 2014 Feb;20(2):130-40. doi: 10.18553/jmcp.2014.20.2.130. PMID 24456314
- [Background] Milsom I, Coyne KS, Nicholson S, Kvasz M, Chen CI, Wein AJ. Global prevalence and economic burden of urgency urinary incontinence: a systematic review. Eur Urol. 2014 Jan;65(1):79-95. doi: 10.1016/j.eururo.2013.08.031. Epub 2013 Aug 27. PMID 24007713
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Onukwugha E, Zuckerman IH, McNally D, Coyne KS, Vats V, Mullins CD. The total economic burden of overactive bladder in the United States: a disease-specific approach. Am J Manag Care. 2009 Mar;15(4 Suppl):S90-7. PMID 19355803
- [Background] Coyne KS, Sexton CC, Bell JA, Thompson CL, Dmochowski R, Bavendam T, Chen CI, Quentin Clemens J. The prevalence of lower urinary tract symptoms (LUTS) and overactive bladder (OAB) by racial/ethnic group and age: results from OAB-POLL. Neurourol Urodyn. 2013 Mar;32(3):230-7. doi: 10.1002/nau.22295. Epub 2012 Jul 27. PMID 22847394